CLINICAL TRIAL: NCT02437617
Title: A Study Exploring the Use of the Foundation Medicine Genomic Profiling Assay in a Phase I Solid Tumor Patient Population
Brief Title: Genomic Profiling Assay in Phase I
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Sponsor
Other Study IDs: PA12-0360
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Advanced Cancers
Keywords: Advanced cancers; Tumor tissue; Genomic profile test; Analysis of treatment outcomes; Molecular profiling; Molecular alteration
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor specimens collected from patients for DNA extraction. All samples residual samples from previously performed biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group #1: Participants who have had tumor molecular analysis performed with the similar clinical characteristics and genomic aberrations but who receive therapy not matched to their aberrations, or who have received results from Foundation Medicine that fail to demonstrate any molecular alteration.
  Interventions: Procedure: Tumor Tissue
- Control Group #2: Participants from historical archives of MD Anderson, no older than two years, who received therapy not matched to their aberrations and are matched not only on the basis of the clinical characteristics, but also, as much as possible, on the basis of genomic aberrations.
  Interventions: Procedure: Tumor Tissue
- Matched Targeted Therapy Group: Participants with tumor aberrations who received matched targeted therapy.

INTERVENTIONS:
Procedure: Tumor Tissue — Tumor tissue collected previously from surgery or a prior biopsy (archived tissue) used for genetic testing.
  Groups: Control Group #1; Control Group #2

SUMMARY:
The goal of this research study is to collect and test tumor tissue from patients with advanced cancers that may be enrolled in Phase 1 studies or other treatments. Researchers will study if the results from genetic testing can help researchers determine which therapy may prove more beneficial for a patient in the future.

DETAILED DESCRIPTION:
If you agree to take part in this study, your tumor tissue collected previously from surgery or a prior biopsy (archived tissue) will be used for genetic testing. Genetic testing looks at whether specific genes are changed (mutated) in the tumor.

The results of the genetic testing will be documented in your medical record. Your doctor may use the results of the genetic testing to help decide which treatment you will have. While awaiting results of the genomic profile assay, you may be enrolled in another treatment either at MD Anderson or near your home. This will be decided by your treating physician.

Your samples will be given a code number when they are sent for genetic testing to Foundation Medicine. No identifying information will be directly linked to your samples. Only the researcher in charge of sending all tissue for testing will have access to the code numbers and be able to link the samples to you. This is to allow medical data related to the samples to be updated as needed. Foundation Medicine will not be able to link this data to you.

Researchers will also review your medical history from before and following the collection of tissue, to learn if the use of genetic testing had any effect on the outcome of your treatment.

This is an investigational study.

Up to 300 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria

1. Patients with advanced cancer.
2. Consent for use of archival tissue from primary or metastatic cancer diagnosis. Note: Patients may currently be enrolled in other investigational protocol including treatment protocols.
3. Control Group #2 only: Control Group #2 will consist of 100 patients from MDACC/Phase I historical archives. Patients (cases no older than 2 years) will be selected based on clinical characteristics and genomic alterations similar to matched targeted therapy group.
4. Patients may have received prior 'matched' therapies; however, at the time of enrollment, patients may not currently be on a known 'matched' therapy, and may not have received a 'matched' therapy as the last treatment if not receiving treatment at the time of consent.
5. Patients who have a life expectancy of greater than 3 months.

Exclusion Criteria:

1. Patients with advanced cancer who are NOT likely to meet the additional enrollment criteria in matched targeted therapy protocols or treatments.
2. Patients who do not have archival tissue available.
3. Patients are excluded if their last treatment before enrollment included a targeted agent matched to a genomic alteration in the patient's tumor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants from MDACC/Phase I historical archives, and participants actively on MDACC/Phase I studies.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-07-13 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Response Rate | 6 months
  Response rate of each of the three cohorts (matched targeted therapy group, control group #1 and control group #2) calculated along with its 95% confidence interval. Response rate defined as proportion of participants who experience complete response (CR) or partial response (PR). Clinical response evaluated according to the RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wheler JJ, Janku F, Naing A, Li Y, Stephen B, Zinner R, Subbiah V, Fu S, Karp D, Falchook GS, Tsimberidou AM, Piha-Paul S, Anderson R, Ke D, Miller V, Yelensky R, Lee JJ, Hong DS, Kurzrock R. Cancer Therapy Directed by Comprehensive Genomic Profiling: A Single Center Study. Cancer Res. 2016 Jul 1;76(13):3690-701. doi: 10.1158/0008-5472.CAN-15-3043. Epub 2016 May 18. PMID 27197177
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org